CLINICAL TRIAL: NCT00538460
Title: Dual-Source CT and STress Cardiac Magnetic Resonance Assessment in the Triage of Patients With Suspected Acute Coronary Syndromes (D-STAT)
Brief Title: Evaluate the Effectiveness and Cost of Stress Cardiac Magnetic Resonance Imaging (MRI) for Non-invasive Evaluation of Lesions Discovered on Computed Tomography Angiography (CCTA)
Acronym: DSTAT
Status: Terminated | Type: Observational
Why Stopped: Lack of staff and funding.
Sponsor: Corewell Health East (Other)
Responsible Party: Kavitha Chinnaiyan, MD, William Beaumont Hospital-Royal Oak, MI
Other Study IDs: 2007-085
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Disease
Keywords: tomography; coronary artery disease; magnetic resonance imaging
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is designed to evaluate the effectiveness and measurable cost impact of stress cardiac MRI for non-invasive evaluation of intermediate lesions discovered on CCTA in low-to-intermediate risk patients admitted to the ED with suspected ACS. Our primary objective is to determine if the strategy of CTA + stress CMR will reduce the length of time in the ED required to establish a definitive diagnosis, compared to CTA + stress MPI.

DETAILED DESCRIPTION:
Non-invasive evaluation of coronary anatomy via multi-slice computed tomography with coronary CT angiography (CCTA) has been shown to provide rapid and accurate non-invasive coronary angiography. Although CCTA can be rapidly and safely performed and despite improving our ability to image coronary arteries in this noninvasive fashion, the limitation of CCTA is lack of physiological information in intermediate lesions, i.e., if a patient has a blockage of 40-60% on CCTA in an artery, it is not possible to know if this is what causes symptoms in a patient. This limitation is currently being overcome by stress testing, commonly with perfusion imaging (nuclear stress test). However, disadvantages of nuclear stress testing include long testing times (usually > 4 hours) and use of radiation. Patients with intermediate/uninterpretable lesions on CCTA will be randomized to MPI or MRI.

The endpoints of the study are:

Primary outcome variables:

1. Length of ED stay until definitive diagnosis (time from ED triage until definitive diagnosis).

Secondary outcome variables will include:

1. Cost of care of an early diagnostic strategy utilizing stress CMR vs. standard care (costs incurred during index hospitalization and 30 day follow up period) in patients with intermediate lesions of CTA.
2. Accuracy of CTA + stress CMR in prediction of occurrence of major adverse cardiac events (MACE) during a 3 month follow-up period, compared to the standard care (CTA + stress/rest MPI): cardiac death, acute myocardial infarction, need for coronary artery revascularization, need for admission or treatment for documented CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chest pain or other symptoms suggestive of acute cardiac ischemia.
2. Low risk TIMI risk score (ie. ≤3)
3. Able to provide informed consent
4. Age equal to or greater than 18 years.

Exclusion Criteria:

1. Electrocardiographic evidence of ischemia, including acute STEMI (ST elevation equal to or greater than 1mm in two or more leads), ST segment depression and/or T wave inversion (not known to be old), or attending physician clinical decision for immediate invasive evaluation.
2. Positive cardiac biomarkers (troponin, myoglobin, and/or creatinine phosphokinase MB fraction).
3. Presence of pre-existing CAD (prior myocardial infarction, prior angiographic evidence of significant CAD, prior coronary bypass surgery) or cardiomyopathy (ejection fraction < 45%)
4. Renal insufficiency (creatinine ≥1.6) or renal failure requiring dialysis.
5. Atrial fibrillation or other markedly irregular rhythm.
6. Inability or refusal to provide informed consent.
7. Psychological unsuitability or extreme claustrophobia.
8. Pregnancy or unknown pregnancy status.
9. Age less than 18 years.
10. Clinical instability as deemed by the attending physician; including cardiogenic shock, hypotension (systolic blood pressure < 90 mmHg), refractory hypertension (systolic blood pressure > 180 mmHg), sustained ventricular or atrial arrhythmia requiring intravenous medications.
11. Patients with known allergy to iodine or shellfish.
12. Inability to tolerate beta blockers, including those with COPD or asthma requiring maintenance inhaled bronchodilators or steroids, complete heart block, second-degree atrioventricular block.
13. Computed tomography imaging, or contrast administration, within the past 48 hours.
14. Use of Viagra or Cialis in the past 24 hours.
15. Patients with known allergy to gadolinium, x-ray dye, Persantine
16. Extreme claustrophobia.
17. Patients with metal implants that prevent MRI scanning
18. Patients with a body weight > 400 lbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers over 18 years of age; both genders
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kavitha Chinnaiyan, MD, Principal Investigator — Corewell Health East; Gilbert Raff, MD, Study Director — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States